CLINICAL TRIAL: NCT04787276
Title: Probiotic E.Coli Nissle 1917 Comparing to Lactulose and Rifaximin in Patients With Mild (Stage 1-2) or Minimal Hepatic Encephalopathy
Brief Title: Efficacy and Safety of E.Coli Nissle 1917 in Patients With Mild (Stage 1-2) or Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Nazarii Kobyliak, Associate Professor, Endocrinology Department, Bogomolets National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HepEN
Record Dates: First submitted 2021-03-02; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis; End Stage Liver DIsease
Keywords: hepatic encephalopathy; Liver Cirrhosis; End Stage Liver DIsease; E.coli Nissle 1917; Probiotic; lactulose; rifaximin
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; End Stage Liver Disease | interventions — Lactulose; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E.coli Nissle 1917 (Experimental): probiotic, oral, for the first 4 days, 1 capsule, and then 2 capsules per day for 1 month treatment
  Interventions: Dietary Supplement: E.coli Nissle 1917
- Lactulose (Active Comparator): will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passed 2-3 semisoft stools per day, 1 months of treatment
  Interventions: Drug: Lactulose
- Rifaximin (Active Comparator): rifaximin, oral, 500 mg BID, 1 months of treatment
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Dietary Supplement: E.coli Nissle 1917 — Probiotic contains biomass of E.coli Nissle 1917, 2,5-25·109 colony forming units - CFU/g
  Other Names: MUTAFLOR capsules
  Arms: E.coli Nissle 1917
Drug: Lactulose — will receive 30-60 ml of lactulose in 2 or 3 divided doses so that patient passed 2-3 semisoft stools per day, 1 months of treatment
  Other Names: DUPHALAC
  Arms: Lactulose
Drug: Rifaximin — rifaximin, oral, 500 mg BID, 1 months of treatment
  Other Names: Alfa Normix
  Arms: Rifaximin

SUMMARY:
The purpose of study to assess the short-term efficacy and safety of probiotic E.coli Nissle 1917 strain comparing to lactulose and rifaximin in patients with mild (Stage 1-2) or minimal hepatic encephalopathy

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed on the basis of liver biopsy, liver stiffness measurement or radiological study;
* presence of minimal or mild (Grade 1-2) HE as defined by West Haven criteria;
* two or more documented episodes of HE in the last 6 months, in addition to at least one episode in the last 3 months;
* subject is capable and willing to comply with all study procedures;
* signed inform consent.

Exclusion Criteria:

* history of taking L-ornithine- L -aspartate, zinc, metronidazole, or neomycin, antibiotics, probiotics and yogurt consumption within 6 weeks;
* subject has a history of allergy or intolerance to lactulose and/or rifaximin;
* alcohol intake during the past 6 month or during follow up;
* recent (6 weeks) gastro-intestinal bleed;
* hepato-cellular carcinoma or liver transplantation;
* renal insufficiency;
* significant comorbid illness such as heart or respiratory failure;
* concurrent infection such as spontaneous bacterial peritonitis, pneumonia or urinary tract infection;
* any neurologic diseases such as alzheimer's disease, parkinson's disease and nonhepatic metabolic encephalopathies;
* subject has any condition or circumstance that would, in the opinion of the Investigator, prevent completion of the study or interfere with analysis of study results, including history of noncompliance with treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Stroop test | 1 month
Change in serum ammonia | 1 month

SECONDARY OUTCOMES:
Change in serum inflammatory cytokine | 1 month
  The level of IL-6, IL-8 and INFγ in pg / ml will be assesed
Bacteriology measured in the stool flora by specialized non-culture techniques | 1 month
  The percentage of patients in each group were evaluated and characterized by a decrease below the normal content of symbiotic bacteria Bifidobacterium (less than 107 CFU / g), lactobacilli (less than 107 CFU / d), E.coli with normal properties (less than 106 CFU / d) and increase in content E.coli with altered properties (more than 106 CFU / g), pathogenic enterobacteria (not normally detected) and fungi of the genus Candida (more than 104 CFU / d)

CONTACTS AND LOCATIONS:
Overall Officials: Elina Manzhalii, PhD, Principal Investigator — Bogomolets National Medical University

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180